CLINICAL TRIAL: NCT01668693
Title: The Endometrial Receptivity Array (ERA) as Diagnosis and Personalized Embryo Transfer (pET) as Treatment in Patients With Receptive Implantation Failure (RIF).
Brief Title: ERA Test in Patients With Recurrent Implantation Failure
Acronym: ERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, MD PhD, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 0600-E-905-JH
Record Dates: First submitted 2012-08-13; First posted 2012-08-20 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Repetitive Implantation Failure
Keywords: Endometrial receptivity; recurrent implantation failure; predictor tool; ERA; customized microarray; personalized embryo transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIF ERA Receptive 1 (Active Comparator): With the "receptive" results from the first Endometrial Receptivity Array (ERA), the patients will undergo embryo transfer on Day 5 of Progesterone administration in the cycle following the ERA diagnosis.
  Interventions: Other: ERA (Endometrial Receptivity Array); Other: Personalized Embryo Transfer
- RIF ERA Non Receptive (Experimental): The "Non Receptive" results of the ERA diagnotic tool will indicate how many more days of Progesterone are necesary in order to obtain the "Receptive" daignosis. A second ERA will take place to confirm receptivity and in the following cycle, the personalized embryo transfer will take place on the day predicted by this diagnostic tool.
  Interventions: Other: ERA (Endometrial Receptivity Array); Other: Personalized Embryo Transfer; Other: Second ERA

INTERVENTIONS:
Other: ERA (Endometrial Receptivity Array) — The diagnostic tool ERA will be performed on all of the patients in order to allocate them in the group "Receptive" or "Non Receptive" and to predict the number of days of Progesterone administration necesary to obtain the "Receptive" prediction.
Other: Personalized Embryo Transfer — When the ERA indicates receptivity, the patient will undergo the embryo transfer on the day indicated by the diagnostic tool.
Other: Second ERA — A second ERA will be performed to confirm receptivity after further administration of Progesterone.
  Arms: RIF ERA Non Receptive

SUMMARY:
The purpose of this study is to demonstrate the clinical efficiency of the Endometrial Receptivity Array (ERA) diagnostic tool in patients with repetitive implantation failure (RIF), leading to the new concept of the personalized window of implantation (pWOI) as diagnostic and treatment of patients with RIF of endometrial origin.

DETAILED DESCRIPTION:
Intervention(s): Endometrial sampling, either at LH+7 in a natural cycle or after 5 days of progesterone in a hormonal replacement cycle (HRT) and personalized embryo transfer (pET) on the designated day guided by the ERA prediction.

Repeated implantation failure (RIF) is an unsolved not well characterized major cause of infertility in otherwise healthy women. Although various definitions of RIF exist, the clinical community agrees that after failure of three IVF cycles, in which one to two morphologically high-grade embryos have been transferred, special protocols must be enforced, although no hard data from RCTs demonstrates that any of the current approaches in RIF have a significant clinical value .

Based on the large amount of information generated about the regulation and deregulation of the genes implicated in the endometrial window of receptivity (WOR), our group has developed a molecular diagnostic tool based on the specific transcriptomic signature that identifies the receptive endometrium at LH+7 in a natural cycle or on day 5 of progesterone impregnation (P+5) after proper estradiol priming in a hormonal replacement therapy (HRT) cycle. The endometrial receptivity array (ERA) consists of a customized array containing 238 genes differentially expressed that is coupled to a computational predictor able to diagnose the personalized endometrial WOI of a given patient, regardless of its histological appearance. The accuracy of the diagnostic tool ERA has been demonstrated to be superior to endometrial histology and results are completely reproducible 29 to 40 months later.

Compelling evidence indicates the existence of an endometrial receptivity alteration in patients with RIF.

The aim of this study is to demonstrate the diagnostic efficiency of the ERA test in RIF patients by identifying putative alterations related to the displacement of their personalized window of receptivity, and the therapeutic implications through personalization of the day of embryo transfer (pET), following the diagnosis obtained by this molecular diagnostic tool. An endometrial biopsy on day LH+7 in a natural cycle or on day P+5 in an HRT cycle and ERA diagnosis of receptive or non-receptive is informed. In receptive cases, embryo transfer (ET) will be performed in subsequent cycles on the indicated day. In non-receptive ERA, the test is to be repeated on the dayindicated by the predictor, and personalized ET guided in subsequent cycles according to ERA diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Women ≤38 years old
* Normal ovarian reserve
* FSH <8mIU/mL
* Cycle with ≥6 MII oocytes/oocyte retrieval
* ≥3 implantation failures in previous IVF/ICSI cycles with transfer of atleast two good quality embryos in each cycle Inclusion Criteria for ovum donation recipients
* ≥3 implantation failures with transfer of atleast two good quality embryos in each cycle
* Endometrial thickness ≥ 6 mm
* Trilaminar pattern after proper progesterone priming

Exclusion Criteria:

* Existance of hydrosalpinx
* Atrophic endometrium < 6 mm
* Previous ectopic or uterine miscarriages
* Presence of myomas or polyps
* Previous embryo transfer with high difficulty and/or bleeding

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Detection of the Receptive or Non Receptive endometrial status according to the ERA test. | 1 months

SECONDARY OUTCOMES:
Pregnancy | 6 weeks
Implantation | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simón, MD PhD, Principal Investigator — ºIGENOMIX / IVI Valencia
Locations (1):
- IVI, Valencia, VAencia, Spain